CLINICAL TRIAL: NCT06590064
Title: The Relationship Between Upper and Lower Extremity Blood Pressure in Thyroid Surgery Patients Under General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Ilsan Cha hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jee Young Lee, Assistant professor, CHA University
Other Study IDs: ICICC-OS-24-02
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Blood Pressure; Diseases of the Thyroid Gland
Keywords: General anesthesia; Thyroid surgery; Lower extremity blood pressure
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group T: Thyroid surgery patients under general anesthesia
  Interventions: Device: Non-invasive Blood Pressure Measurement

INTERVENTIONS:
Device: Non-invasive Blood Pressure Measurement — Non-invasive Blood Pressure Measurement in Both Upper and Lower Limbs

SUMMARY:
The goal of this observational study is to clarify the relationship between upper and lower limb blood pressure in thyroid surgery patients under general anesthesia. The hemodynamic state during anesthesia is different from that during the awake state. Therefore, to assess whether the difference in blood pressure between the upper and lower limbs observed in the awake state is consistent with that observed under general anesthesia, the investigators will compare the inter-limb blood pressure differences before anesthesia induction and during general anesthesia.

DETAILED DESCRIPTION:
Non-invasive blood pressure measurement during surgery is typically conducted on the upper arm, and previous studies about the relationship between intraoperative blood pressure fluctuation and postoperative mortality and morbility have also based on the upper arm measurements. However, in clinical practice, if monitoring blood pressure in the upper arm is not feasible during surgery, the cuff usually be placed on the ankle.

According to a previous study, the systolic blood pressure at the ankle is approximately 17.0 mmHg higher than the systolic blood pressure at the arm in the supine position (95% CI 15.4-21.3 mmHg), while the diastolic blood pressure did not show significant differences in awake state. Since the hemodynamic state of patients under anesthesia differs from that of awake patients, there is insufficient evidence to directly apply the known differences between upper and lower limb blood pressures in awake patients to set target blood pressure ranges during anesthesia. As a result, anesthesiologists often rely on clinical judgment in these situations.

Therefore, this study sets the null hypothesis that 'the differences in blood pressure between the upper and lower limbs before and after anesthesia are the same.' The goal is to determine whether the previously known relationship between upper and lower limb blood pressures in awake patients can be applied to patients under general anesthesia. Additionally, this study aims to investigate the relationship between upper and lower limb blood pressures when the lower limb blood pressure is outside the normal range during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients having elective thyroid surgery under general anesthesia
* Aged between 20 to 80 years old
* American Society of Anesthesiologist(ASA) Physical Status Class I or II
* Individuals who have voluntarily given written consent to participate in this clinical study

Exclusion Criteria:

* Patients with Diabetes Mellitus or Peripheral vascular disease
* Patients with a history of Heart disease; Myocardial infarction, Heart failure, etc.
* Patients with Arrhythmia
* Patients with musculoskeletal abnormalities
* Patients for whom the placement of a non-invasive blood pressure cuff is contraindicated: inflammatory diseases or wounds causing pain at the cuff site, severe edema, thrombophlebitis, etc.
* Other cases deemed unsuitable for the study by the researcher: absence of appropriately sized blood pressure cuffs, placement of a pressurized blood pressure cuff expected to affect the induction and maintenance of general anesthesia, history of mental illness, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving elective thyroid surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
d_MBP(awake) | Simultaneously measured values in operating room before anesthesia induction
  Difference between upper and lower extremities mean blood pressure in awake state
d_MBP(GA) | Simultaneously measured values during general anesthesia in a stable state without significant stimulation
  Difference between upper and lower extremities mean blood pressure during general anesthesia

SECONDARY OUTCOMES:
d_SBP(awake) | Simultaneously measured values in operating room before anesthesia induction
  Difference between upper and lower extremities systolic blood pressure in awake state
d_SBP(GA) | Simultaneously measured values during general anesthesia in a stable state without significant stimulation
  Difference between upper and lower extremities systolic blood pressure during general anesthesia
d_DBP(awake) | Simultaneously measured values in operating room before anesthesia induction
  Difference between upper and lower extremities diastolic blood pressure in awake state
d_DBP(GA) | Simultaneously measured values during general anesthesia in a stable state without significant stimulation
  Difference between upper and lower extremities diastolic blood pressure during general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: JOOHYUN LEE, Principal Investigator — Department of Anesthesia and Pain medicine, Ilsan Cha hospital
Locations (1):
- Ilsan Cha hospital, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Sheppard JP, Albasri A, Franssen M, Fletcher B, Pealing L, Roberts N, Obeid A, Pucci M, McManus RJ, Martin U; British and Irish Hypertension Society. Defining the relationship between arm and leg blood pressure readings: a systematic review and meta-analysis. J Hypertens. 2019 Apr;37(4):660-670. doi: 10.1097/HJH.0000000000001958. PMID 30817444
- [Background] Jessen MK, Vallentin MF, Holmberg MJ, Bolther M, Hansen FB, Holst JM, Magnussen A, Hansen NS, Johannsen CM, Enevoldsen J, Jensen TH, Roessler LL, Lind PC, Klitholm MP, Eggertsen MA, Caap P, Boye C, Dabrowski KM, Vormfenne L, Hoybye M, Henriksen J, Karlsson CM, Balleby IR, Rasmussen MS, Paelestik K, Granfeldt A, Andersen LW. Goal-directed haemodynamic therapy during general anaesthesia for noncardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2022 Mar;128(3):416-433. doi: 10.1016/j.bja.2021.10.046. Epub 2021 Dec 13. PMID 34916049